CLINICAL TRIAL: NCT04553458
Title: Factors Affecting Post-treatment Outcomes in Patients With Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Emad Ali Ahmed Ali, Principal investigator, Sohag University
Other Study IDs: 22/09/2020
Record Dates: First submitted 2020-09-05; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; HCC; Hepatoma; primary liver tumours
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation; Hepatectomy; Ethanol; Neoadjuvant Therapy; Sorafenib; Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Favorable outcome: Cure or stable disease
  Interventions: Device: Radiofrequency ablation; Drug: Trance-arterial chemoembolization; Procedure: Liver resection; Combination Product: Combined radiofrequency ablation + percutaneous ethanol injection; Drug: Percutaneous ethanol injection
- Unfavorable outcome: Progressive (deteriorate/Recurrence) or Death
  Interventions: Device: Radiofrequency ablation; Drug: Trance-arterial chemoembolization; Combination Product: Combined radiofrequency ablation + percutaneous ethanol injection; Drug: Percutaneous ethanol injection; Drug: Systemic chemotherapy; Drug: Sorafenib; Dietary Supplement: Viscum; Drug: Symptomatic treatment

INTERVENTIONS:
Device: Radiofrequency ablation — Radiofrequency ablation of the tumour
Drug: Trance-arterial chemoembolization — Trance-arterial chemotherapy
  Other Names: transcatheter arterial chemoembolization
Procedure: Liver resection — non-anatomical or anatomical liver resection
  Groups: Favorable outcome
Combination Product: Combined radiofrequency ablation + percutaneous ethanol injection — combined therapy
Drug: Percutaneous ethanol injection — Percutaneous ethanol injection of HCC
  Other Names: ETHANOL
Drug: Systemic chemotherapy — Systemic chemotherapy
  Other Names: MIXED
  Groups: Unfavorable outcome
Drug: Sorafenib — Sorafenib
  Other Names: NEXAVAR
  Groups: Unfavorable outcome
Dietary Supplement: Viscum — Viscum for HCC
  Groups: Unfavorable outcome
Drug: Symptomatic treatment — Symptomatic treatment
  Other Names: SUPPORTIVE
  Groups: Unfavorable outcome

SUMMARY:
EASL and mRECIST criteria differ from each other in terms of the number of target lesions (all versus < = 2) and calculation method (bidimensional versus unidimensional). Therefore, the investigators aimed to retrospectively analyze and compare the clinical outcomes among patients with hepatocellular carcinoma who were treated with different modalities of therapy according to the BCLC classification, and detect the possible predictors of post-treatment outcomes.

DETAILED DESCRIPTION:
Background:

EASL and mRECIST criteria differ from each other in terms of the number of target lesions (all versus < = 2) and calculation method (bidimensional versus unidimensional). Therefore, the investigators aimed to retrospectively analyze and compare the clinical outcomes among patients with hepatocellular carcinoma (HCC) who were treated with different modalities of therapy according to the BCLC classification, and detect the possible predictors of post-treatment outcomes.

Methods:

This work was conducted at the departments of tropical medicine and gastroenterology, internal medicine, and general surgery. This study included patients that matched our eligibility criteria for a period of five years started from June 2015 to May 2020. The study purpose was to retrospectively analyze the clinical outcomes among patients with HCC who were treated with different modalities of therapy according to the BCLC classification, and detect the possible predictors of post-treatment favorable outcomes. The data of the patients were extracted and retrospectively reviewed from the patients' records and the databases of both hospitals (SUH and SOI).

During the period of recruitment, 407 patients diagnosed with HCC admitted to our departments and followed-up attending outpatient clinics, Sohag University Hospitals, over a 5 years period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* with hepatocellular carcinoma

Exclusion Criteria:

* severely-ill patients
* With other system comorbidities,
* presence of extrahepatic metastasis,
* patients who dropped from the follow-up list after treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This work was conducted at the departments of tropical medicine and gastroenterology, internal medicine, and general surgery. This study included patients that matched our eligibility criteria for a period of five years started from June 2015 to May 2020. The study purpose was to retrospectively analyze the clinical outcomes among patients with HCC who were treated with different modalities of therapy according to the BCLC classification, and detect the possible predictors of post-treatment favorable outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
CURE (Number of patients cured completely from the disease) | one-year
  the HCC is treated (disappearance of all lesions)
STABLE Disease (Number of patients with neither progression nor cure from the disease) | one-year
  NONE of the other outcomes' criteria
PROGRESSIVE((Number of patients with progression of the disease) (measured by follow-up CT scans, increase in size, appearance of new intratumoral lesions, or appearance of new lesions | one-year
  increase in size - appearance of new intratumoral lesions - new lesions

SECONDARY OUTCOMES:
DEATH (Number of patients died from the disease) | one-year
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Emad A. Ahmed, MD, PhD, Principal Investigator — Sohag University